CLINICAL TRIAL: NCT04949256
Title: A Phase 3, Randomized Study to Evaluate the Efficacy and Safety of Pembrolizumab (MK-3475) + Lenvatinib (E7080/MK-7902) + Chemotherapy Compared With Standard of Care as First-line Intervention in Participants With Metastatic Esophageal Carcinoma
Brief Title: Efficacy and Safety of Pembrolizumab (MK-3475) Plus Lenvatinib (E7080/MK-7902) Plus Chemotherapy in Participants With Metastatic Esophageal Carcinoma (MK-7902-014/E7080-G000-320/LEAP-014)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7902-014; MK-7902-014 (Other: MSD); LEAP-014 (Other: MSD); E7080-G000-320 (Other: Eisai); U1111-1280-1020 (Registry Identifier: UTN); 2022-501342-29-00 (Registry Identifier: EU CT); 2020-001911-26 (EudraCT Number)
Record Dates: First submitted 2021-06-29; First posted 2021-07-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Esophageal Squamous Cell Carcinoma
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib; Cisplatin; Fluorouracil; Oxaliplatin; Leucovorin; Levoleucovorin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Pembrolizumab + Lenvatinib + Chemotherapy (Experimental): In the Induction phase, participants receive pembrolizumab 400mg intravenously (IV) every 6 weeks (Q6W) for 2 cycles (each cycle length = 6 weeks) plus Lenvatinib 8 mg orally (PO) once daily (QD) plus chemotherapy with FP (cisplatin 80 mg/m^2 and 5-FU 400 mg/m^2 followed by 2400 mg/m^2) or TP (paclitaxel 175 mg/m^2 and cisplatin 75 mg/m^2) IV every 3 weeks for 4 administrations at the investigator's discretion (approximately 12 weeks). In the Consolidation phase, participants receive pembrolizumab 400 mg IV Q6W for 16 cycles (each cycle length = 6 weeks) and Lenvatinib 20 mg PO until progressive disease or discontinuation (approximately 96 weeks).
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib; Drug: Cisplatin; Drug: 5-FU; Drug: Paclitaxel
- Part 2: Pembrolizumab + Lenvatinib + Chemotherapy (Experimental): In the Induction phase, participants receive pembrolizumab 400mg intravenously (IV) every 6 weeks (Q6W) for 2 cycles (each cycle length = 6 weeks) plus Lenvatinib 8 mg orally (PO) once daily (QD) plus chemotherapy with FP (cisplatin 80 mg/m^2 and 5-FU 4000 mg/m^2) or TP (paclitaxel 175 mg/m^2 and cisplatin 75 mg/m^2) IV every 3 weeks for 4 administrations or mFOLFOX6 (oxaliplatin 85 mg/m^2, 5-FU 400 mg/m^2 followed by 2400 mg/m^2, and leucovorin 400 mg/m^2 [or levoleucovorin 200 mg/m^2] once every 2 weeks [Q2W] for 6 administrations at the investigator's discretion (approximately 12 weeks). In the Consolidation phase, participants receive pembrolizumab 400 mg IV Q6W for 16 cycles (each cycle length = 6 weeks) and Lenvatinib 20 mg PO until progressive disease or discontinuation (approximately 96 weeks).
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib; Drug: Cisplatin; Drug: 5-FU; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Levoleucovorin; Drug: Paclitaxel
- Part 2: Pembrolizumab + Chemotherapy (Active Comparator): Participants receive pembrolizumab 400 mg IV every 6 weeks for 18 cycles (each cycle length = 6 weeks, approximately 2 years) plus chemotherapy with FP (cisplatin 80 mg/m^2 IV Q3W for up to 6 administrations [up to ~18 weeks] and 5-FU 4000 mg/m^2 IV Q3W for up to 35 administrations [up to ~2 years]) or TP (paclitaxel 175 mg/m^2 and cisplatin 75 mg/m^2 Q3W for up 6 administrations [up to ~18 weeks]) or in combination with mFOLFOX6 (oxaliplatin 85 mg/m^2, 5-FU 400 mg/m^2 followed by 2400 mg/m^2 and leucovorin 400 mg/m^2 [or levoleucovorin 200 mg/m^2] IV Q2W for up to 52 administrations [approximately 2 years]).
  Interventions: Biological: Pembrolizumab; Drug: 5-FU; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Levoleucovorin; Drug: Paclitaxel

INTERVENTIONS:
Biological: Pembrolizumab — 400 mg once every 6-week-cycle, via IV infusion.
  Other Names: MK-3475; KEYTRUDA®
Drug: Lenvatinib — 8 mg QD (Induction) or 20 mg QD (Consolidation) via oral capsule.
  Other Names: MK-7902; E7080; LENVIMA®
  Arms: Part 1: Pembrolizumab + Lenvatinib + Chemotherapy; Part 2: Pembrolizumab + Lenvatinib + Chemotherapy
Drug: Cisplatin — 80 mg/m^2 Q3W via IV infusion, as part of investigator's choice FP chemotherapy or 75 mg/m^2 Q3W via infusion, as part of investigator's choice TP chemotherapy.
  Other Names: PLATINOL®
  Arms: Part 1: Pembrolizumab + Lenvatinib + Chemotherapy; Part 2: Pembrolizumab + Lenvatinib + Chemotherapy
Drug: 5-FU — 4000 mg/m^2 Q3W via IV infusion, as part of investigator's choice FP chemotherapy or 400 mg/m^2 Q2W via bolus IV infusion followed by 2400 mg/m^2 Q2W via continuous IV infusion, as part of investigator's choice mFOLFOX6 chemotherapy.
  Other Names: ADRUCIL®
Drug: Oxaliplatin — 85 mg/m^2 Q2W via IV infusion, as part of investigator's choice mFOLFOX6 chemotherapy.
  Other Names: ELOXATIN®
  Arms: Part 2: Pembrolizumab + Chemotherapy; Part 2: Pembrolizumab + Lenvatinib + Chemotherapy
Drug: Leucovorin — 400 mg/m^2 Q2W as part of investigator's choice mFOLFOX6 chemotherapy.
  Other Names: calcium folinate; folinic acid; WELLCOVORIN®
  Arms: Part 2: Pembrolizumab + Chemotherapy; Part 2: Pembrolizumab + Lenvatinib + Chemotherapy
Drug: Levoleucovorin — 200 mg/m^2 Q2W as part of investigator's choice mFOLFOX6 chemotherapy.
  Other Names: calcium levofolinate; levofolinic acid; FUSILEV®
  Arms: Part 2: Pembrolizumab + Chemotherapy; Part 2: Pembrolizumab + Lenvatinib + Chemotherapy
Drug: Paclitaxel — 175 mg/m^2 Q3W via IV infusion, as part of investigator's choice TP chemotherapy.
  Other Names: TAXOL®; ONXAL®

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pembrolizumab plus lenvatinib plus chemotherapy compared with pembrolizumab plus chemotherapy as first-line intervention in participants with metastatic esophageal carcinoma.

The primary hypotheses are that pembrolizumab plus lenvatinib plus chemotherapy is superior to pembrolizumab plus chemotherapy with respect to overall survival (OS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by blinded independent central review (BICR).

As of Amendment 09, Study MK-7902-014 will begin close out activities. Any participant who discontinues study intervention for any reason will be discontinued from the study without further follow-up. Second Course and treatment beyond disease progression will no longer be offered. No safety concerns contributed to the termination of this study.

DETAILED DESCRIPTION:
There will be 2 parts to the study: the cisplatin and 5-fluorouracil (5-FU) (FP) and paclitaxel and cisplatin (TP) Safety Run-in (Part 1) and the Main Study (Part 2). In Part 1 (FP and TP Safety Run-in), participants will be treated with pembrolizumab plus lenvatinib plus FP or TP. Dose-limiting toxicities, safety, and tolerability will be assessed.

In Part 2 (Main Study), participants (not including those participating in Part 1) will be treated with pembrolizumab plus lenvatinib plus chemotherapy or pembrolizumab plus chemotherapy. Efficacy, safety, and tolerability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of metastatic squamous cell carcinoma of the esophagus
* Male participants are abstinent from heterosexual intercourse or agree to use contraception during the intervention period and for at least 7 days after the last dose of lenvatinib or 90 days after the last dose of chemotherapy, whichever comes last; 7 days after lenvatinib is stopped, if the participant is on pembrolizumab only and is greater than 90 days post chemotherapy, no male contraception is needed
* Female participant is not pregnant or breastfeeding and is not a woman of childbearing potential (WOCBP) or is a WOCBP using a contraceptive method that is highly effective or is abstinent from heterosexual intercourse as their preferred and usual lifestyle during the intervention period and for at least 120 days after the last dose of pembrolizumab, 30 days after the last dose of lenvatinib, or 180 days after the last dose of chemotherapy, whichever occurs last, and agrees not to donate eggs during this period
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP≤150/90 millimeters of mercury (mm Hg) with no change in antihypertensive medications within 1 week prior to randomization
* Has adequate organ function

Exclusion Criteria:

* Has had previous therapy for locally advanced unresectable or metastatic esophageal cancer
* Has locally advanced esophageal carcinoma
* Has metastatic adenocarcinoma of the esophagus
* Has direct invasion into adjacent organs such as the aorta or trachea
* Has radiographic evidence of encasement of a major blood vessel, or of intratumoral cavitation
* Has perforation risks or significant gastrointestinal (GI) bleeding
* Has had clinically significant hemoptysis within 3 weeks prior to the first dose of study drug or tumor bleeding within 2 weeks prior to the first dose of study intervention
* Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage or medical intervention
* Has GI obstruction, poor oral intake, difficulty in taking oral medication, or existing esophageal stent
* Has had major surgery, open biopsy, or significant traumatic injury within 3 weeks prior to first dose of study interventions
* Has received prior radiotherapy within 2 weeks of start of study intervention or have had a history of radiation pneumonitis
* Has received a live or live attenuated vaccine within 30 days prior to the first dose of study intervention; administration of killed vaccines is allowed
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any form of immunosuppressive therapy within 7 days prior to the first dose of study intervention, or has a history of organ transplant, including allogeneic stem cell transplant
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in past 2 years; replacement therapy is not considered a form of systemic treatment and is allowed
* Has a history of non-infectious pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease
* Has poorly controlled diarrhea
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention
* Has peripheral neuropathy ≥Grade 2
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B or know active Hepatitis C virus infection
* Has a weight loss of >20% within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Part 1 (FP and TP Safety Run-in): Number of Participants With Dose Limiting Toxicities (DLTs) | Up to ~21 days
  Hematologic DLTs are defined as Grade 4 neutropenia lasting for ≥7 days, Grade 3 or Grade 4 febrile neutropenia, Grade 3 thrombocytopenia with bleeding, Grade 4 thrombocytopenia, or Grade 4 anemia. Other nonhematologic toxicities considered a DLT include any other Grade 4 or Grade 5 toxicity, Grade 3 toxicities lasting >3 days (excluding nausea, vomiting, and diarrhea controlled by medical intervention within 72 hours, and Grade 3 rash in the absence of desquamation with no mucosal involvement), Grade 3 hypertension not able to be controlled by medication, ≥Grade 3 gastrointestinal perforation, ≥Grade 3 wound dehiscence requiring medical or surgical intervention, any grade thromboembolic event or any Grade 3 nonhematologic laboratory value requiring medical intervention or hospitalization. The number of participants in Part 1 with DLTs will be presented.
Part 1 (FP and TP Safety Run-in): Number of Participants With Adverse Events (AEs) | Up to ~53 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants in Part 1 with AEs will be presented.
Part 1 (FP and TP Safety Run-in): Number of Participants who Discontinued Study Treatment Due to an AE | Up to ~53 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants in Part 1 who discontinue study treatment due to an AE will be presented.
Part 2 (Main Study): Overall Survival (OS) in all Participants | Up to ~48 months
  OS is defined as the time from randomization to death due to any cause. OS in Part 2 for all randomized participants will be presented.

SECONDARY OUTCOMES:
Part 2 (Main Study): Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in all Participants | Up to ~42 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 by BICR or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. RECIST 1.1 has been adjusted to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ. PFS in Part 2 for all randomized participants will be presented.
Part 2 (Main Study): Objective Response Rate (ORR) per RECIST 1.1 as Assessed by BICR in all Participants | Up to ~42 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions), per RECIST 1.1 adjusted to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, as assessed by BICR. ORR in Part 2 for all randomized participants will be presented.
Part 2 (Main Study): Duration of Response (DOR) per RECIST 1.1 as Assessed by BICR in all Participants | Up to ~42 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions), per RECIST 1.1 by BICR, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. RECIST 1.1 has been adjusted to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ. DOR in Part 2 for all randomized participants will be presented.
Part 2 (Main Study): OS in Participants With Programmed Cell Death-Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥10 | Up to ~48 months
  OS is defined as the time from randomization to death due to any cause. OS in Part 2 for randomized participants with PD-L1 CPS ≥10 will be presented.
Part 2 (Main Study): PFS per RECIST 1.1 as Assessed by BICR in Participants With PD-L1 CPS ≥10 | Up to ~42 months
  PFS is defined as the time from randomization to the first documented PD per RECIST 1.1 by BICR or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. RECIST 1.1 has been adjusted to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ. PFS in Part 2 for randomized participants with PD-L1 CPS ≥10 will be presented.
Part 2 (Main Study): ORR per RECIST 1.1 as Assessed by BICR in Participants With PD-L1 CPS ≥10 | Up to ~42 months
  ORR is defined as the percentage of participants with CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions), per RECIST 1.1 adjusted to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, as assessed by BICR. ORR in Part 2 for randomized participants with PD-L1 CPS ≥10 will be presented.
Part 2 (Main Study): DOR per RECIST 1.1 as Assessed by BICR in Participants With PD-L1 CPS ≥10 | Up to ~42 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions), per RECIST 1.1 by BICR, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. RECIST 1.1 has been adjusted to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ. DOR in Part 2 for randomized participants with PD-L1 CPS ≥10 will be presented.
Part 2 (Main Study): Number of Participants With AEs | Up to ~53 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants in Part 2 with AEs will be presented.
Part 2 (Main Study): Number of Participants who Discontinued Study Treatment Due to an AE | Up to ~53 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants in Part 2 who discontinue study treatment due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (198):
- United States (15):
  - City of Hope ( Site 0102), Duarte, California
  - MedStar Washington Hospital Center ( Site 0186), Washington D.C., District of Columbia
  - James Graham Brown Cancer Center ( Site 0117), Louisville, Kentucky
  - Norton Cancer Institute ( Site 0116), Louisville, Kentucky
  - Johns Hopkins Bayview Medical Center ( Site 0152), Baltimore, Maryland
  - UMASS Memorial Medical Center ( Site 0120), Worcester, Massachusetts
  - Capital Health Medical Center - Hopewell ( Site 0189), Pennington, New Jersey
  - Hematology-Oncology Associates of CNY ( Site 0173), East Syracuse, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0132), New York, New York
  - Weill Cornell Medical College ( Site 0133), New York, New York
  - St. Luke's University Health Network ( Site 0185), Bethlehem, Pennsylvania
  - AHN Allegheny General Hospital ( Site 0164), Pittsburgh, Pennsylvania
  - Medical University of South Carolina-Hollings Cancer Center ( Site 0177), Charleston, South Carolina
  - VCU Health Adult Outpatient Pavillion ( Site 0160), Richmond, Virginia
  - Seattle Cancer Care Alliance ( Site 0145), Seattle, Washington
- Argentina (11):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA ( Site 0203), Berazategui, Buenos Aires
  - IDIM Instituto de Diagnostico e Investigaciones Metabolicas ( Site 0202), CABA, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 0205), Mar del Plata, Buenos Aires
  - Fundacion Estudios Clinicos-Oncology ( Site 0215), Rosario, Santa Fe Province
  - Sanatorio Parque ( Site 0206), Rosario, Santa Fe Province
  - Hospital Provincial del Centenario ( Site 0217), Rosario, Santa Fe Province
  - Fundacion Favaloro ( Site 0201), Buenos Aires
  - Fundación Respirar ( Site 0216), Buenos Aires
  - Hospital Italiano de Córdoba ( Site 0218), Córdoba
  - Fundación CORI para la Investigación y Prevención del Cáncer ( Site 0221), La Rioja
  - Instituto San Marcos ( Site 0213), San Juan
- Canada (3):
  - CancerCare Manitoba ( Site 0001), Winnipeg, Manitoba
  - Princess Margaret Cancer Centre ( Site 0004), Toronto, Ontario
  - Hotel-Dieu de Levis ( Site 0013), Lévis, Quebec
- Chile (6):
  - Fundacion Arturo Lopez Perez FALP ( Site 0403), Santiago, Region M. de Santiago
  - Oncovida ( Site 0413), Santiago, Region M. de Santiago
  - Clínica San Carlos de Apoquindo Red Salud UC Christus ( Site 0407), Santiago, Region M. de Santiago
  - Bradford Hill Centro de Investigaciones Clinicas ( Site 0404), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 0412), Temuco, Región de la Araucanía
  - Centro de Investigacion y desarrollo Oncologico SpA - CIDO SpA ( Site 0401), Temuco, Región de la Araucanía
- China (29):
  - Anhui Provincial Cancer Hospital ( Site 8058), Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University ( Site 8026), Hefei, Anhui
  - Beijing Cancer Hospital ( Site 8001), Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital ( Site 8029), Fuzhou, Fujian
  - Zhongshan Hospital Affiliated to Xiamen University ( Site 8055), Xiamen, Fujian
  - The First Affiliated Hospital of Xiamen University ( Site 8003), Xiamen City, Fujian Province, Fujian
  - The First Affiliated Hospital.Sun Yat-sen University ( Site 8047), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 8031), Guangzhou, Guangdong
  - The Third Xiangya Hospital of Central South University ( Site 8046), Changsha, Hainan
  - The First Affiliated Hospital of Hainan Medical University ( Site 8042), Haikou, Hainan
  - Affiliated Hospital of Chengde Medical Univeristy ( Site 8053), Chengde, Hebei
  - Harbin Medical University Cancer Hospital ( Site 8009), Harbin, Heilongjiang
  - Anyang Cancer Hospital ( Site 8006), Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science &Technology-Tumor ( Site 8036), Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University ( Site 8018), Xinxiang, Henan
  - Tongji Medical College Huazhong Uinversity Of Science and Technology ( Site 8025), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 8014), Wuhan, Hubei
  - Affiliated hospital of Jiangnan university ( Site 8049), Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University ( Site 8015), Xuzhou, Jiangsu
  - Jilin Cancer Hospital ( Site 8016), Changchun, Jilin
  - Jinan Central Hospital ( Site 8052), Jinan, Shandong
  - Shandong Cancer Hospital ( Site 8060), Jinan, Shandong
  - Affiliated Hospital of Jining Medical University ( Site 8017), Jining, Shandong
  - Linyi Cancer Hospital- Medical Oncology Department ( Site 8051), Linyi, Shandong
  - Shanxi Provincial Cancer Hospital ( Site 8019), Taiyuan, Shanxi
  - West China Hospital of Sichuan University ( Site 8048), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital ( Site 8035), Tianjin, Tianjin Municipality
  - The Affiliated Cancer Hospital of Xinjiang Medical University. ( Site 8041), Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital ( Site 8021), Hangzhou, Zhejiang
- Costa Rica (4):
  - ICIMED-Oncology Research Unit ( Site 0903), San José, Provincia de San José
  - PROCLINICAL Pharma ( Site 0904), San José, Provincia de San José
  - CIMCA Centro de Investigacion y Manejo del Cancer ( Site 0902), San José
  - Onco Tech S A ( Site 0901), San José
- Denmark (2):
  - Rigshospitalet ( Site 2102), Copenhagen, Capital Region
  - Odense University Hospital ( Site 2101), Odense, Region Syddanmark
- France (13):
  - Institut De Cancerologie De Lorraine ( Site 1010), Vandœuvre-lès-Nancy, Ain
  - Institut de cancérologie Strasbourg Europe (ICANS) ( Site 1014), Strasbourg, Alsace
  - Centre François Baclesse ( Site 1009), Caen, Calvados
  - Centre Georges Francois Leclerc ( Site 1008), Dijon, Cote-d Or
  - C.H. regional Unv. de Brest - Hopital La Cavale Blanche - Institut de Cancerologie et d Imagerie ( S, Brest, Finistere
  - CHU Besançon ( Site 1015), Besançon, Franche-Comte
  - CHU Bordeaux Haut-Leveque ( Site 1012), Pessac, Gironde
  - Institut du Cancer de Montpellier ( Site 1002), Montpellier, Herault
  - CHRU de Tours - Hopital Bretonneau ( Site 1018), Tours, Indre-et-Loire
  - Institut De Cancerologie De L Ouest ( Site 1003), Saint-Herblain, Loire-Atlantique
  - Hôpital Claude Huriez ( Site 1030), Lille, Nord
  - Hopital Henri Mondor ( Site 1007), Créteil, Val-de-Marne
  - Hopital Saint Louis ( Site 1029), Paris
- Guatemala (4):
  - Centro Regional de Sub Especialidades Medicas SA ( Site 0604), Guatemala, Departamento de Quetzaltenango
  - MEDI-K ( Site 0601), Guatemala City
  - Oncomedica ( Site 0602), Guatemala City
  - Soluciones Gastrointestinales S.A. ( Site 0607), Guatemala City
- Hong Kong (2):
  - Queen Mary Hospital ( Site 4001), Hong Kong
  - Queen Elizabeth Hospital. ( Site 4004), Kowloon
- Hungary (4):
  - Pecsi Tudomanyegyetem AOK ( Site 1204), Pécs, Baranya
  - Petz Aladar Egyetemi Oktato Korhaz ( Site 1210), Győr, Győr-Moson-Sopron
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház ( Site 1203), Szolnok, Jász-Nagykun-Szolnok
  - Orszagos Onkologiai Intezet ( Site 1207), Budapest
- Italy (12):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori-Oncologia Medica ( Site 1313), Meldola, Emilia-Romagna
  - A.O.U. Santa Maria della Misericordia di Udine ( Site 1302), Udine, Friuli Venezia Giulia
  - Humanitas Research Hospital ( Site 1309), Rozzano, Lombardy
  - Azienda Ospedaliera Universitaria Pisana ( Site 1312), Pisa, Tuscany
  - Istituto Oncologico Veneto IRCCS-Oncologia Medica 1 ( Site 1311), Padua, Veneto
  - Azienda Ospedaliera Mater Domini-Translational Oncology Unit ( Site 1314), Catanzaro
  - Azienda Ospedaliero Universitaria Careggi ( Site 1301), Florence
  - IRCCS Ospedale San Raffaele di Milano ( Site 1304), Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 1306), Milan
  - A.O. Universitaria di Modena ( Site 1307), Modena
  - A.O.U. Universita degli Studi della Campania-Luigi Vanvitelli ( Site 1305), Napoli
  - Universita Cattolica del Sacro Cuore - Policlinico Gemelli ( Site 1310), Roma
- Japan (27):
  - Aichi Cancer Center Hospital ( Site 9006), Nagoya, Aichi-ken
  - Chiba Cancer Center ( Site 9023), Chiba, Chiba
  - National Cancer Center Hospital East ( Site 9002), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 9019), Matsuyama, Ehime
  - Hyogo Cancer Center ( Site 9014), Akashi, Hyōgo
  - Ibaraki Prefectural Central Hospital ( Site 9007), Kasama, Ibaraki
  - Kagawa University Hospital ( Site 9015), Kita-gun, Kagawa-ken
  - Kanagawa Cancer Center ( Site 9004), Yokohama, Kanagawa
  - Tohoku University Hospital ( Site 9013), Sendai, Miyagi
  - Niigata Cancer Center Hospital ( Site 9022), Niigata, Niigata
  - Kindai University Hospital ( Site 9017), Sayama, Osaka
  - Osaka University Hospital ( Site 9021), Suita, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 9008), Takatsuki, Osaka
  - Saitama Prefectural Cancer Center ( Site 9003), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center ( Site 9016), Nakatogari, Shizuoka
  - Tokyo Metropolitan Komagome Hospital ( Site 9028), Bunkyo Ku, Tokyo
  - Toranomon Hospital ( Site 9026), Minato-ku, Tokyo
  - Showa University Hospital ( Site 9025), Shinagawa, Tokyo
  - National Hospital Organization Kyushu Cancer Center ( Site 9010), Fukuoka
  - University Hospital,Kyoto Prefectural University of Medicine ( Site 9027), Kyoto
  - Kyoto University Hospital ( Site 9011), Kyoto
  - Okayama University Hospital ( Site 9024), Okayama
  - Osaka International Cancer Institute ( Site 9009), Osaka
  - Osaka General Medical Center ( Site 9018), Osaka
  - National Cancer Center Hospital ( Site 9001), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 9005), Tokyo
  - Keio University Hospital ( Site 9020), Tokyo
- Malaysia (3):
  - University Malaya Medical Centre ( Site 9101), Lembah Pantai, Kuala Lumpur
  - Sarawak General Hospital-Radiotherapy Unit ( Site 9100), Kuching, Sarawak
  - Hospital Kuala Lumpur ( Site 9104), Kuala Lumpur
- Romania (6):
  - MEMORIAL HEALTHCARE INTERNATIONAL S.R.L. ( Site 2201), Bucharest, București
  - Cardiomed SRL Cluj-Napoca-Medical Oncology ( Site 2207), Cluj-Napoca, Cluj
  - SC Radiotherapy Center Cluj SRL ( Site 2202), Comuna Floresti, Cluj
  - Ovidius Clinical Hospital OCH-Oncology and Hematology ( Site 2203), Ovidiu, Constanța County
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 2204), Craiova, Dolj
  - Policlinica Oncomed SRL ( Site 2206), Timișoara, Timiș County
- Russia (7):
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 1507), Ufa, Baskortostan, Respublika
  - GBUZ LOKB ( Site 1502), Saint-Petersburg, Leningradskaya Oblast'
  - FSBI National Medical Oncology Research Center n.a. N.N. Blokhina ( Site 1510), Moscow, Moscow
  - Academician I.P. Pavlov First St. Petersburg State Medical University ( Site 1519), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 1503), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH named after professor M.Z. Sigal ( Site 150, Kazan', Tatarstan, Respublika
  - SAIH of Tyumen reg "Multifield clinical medical center "Medical city" ( Site 1520), Tyumen, Tyumen Oblast
- National Cancer Centre Singapore ( Site 9201), Singapore, Central Singapore, Singapore
- South Africa (2):
  - Wits Clinical Research ( Site 9502), Johannesburg, Gauteng
  - The Oncology Centre ( Site 9505), Durban, KwaZulu-Natal
- South Korea (5):
  - Seoul National University Bundang Hospital ( Site 5006), Seongnam-si, Kyonggi-do
  - Asan Medical Center ( Site 5002), Songpagu, Seoul
  - Severance Hospital ( Site 5003), Seoul
  - Samsung Medical Center ( Site 5005), Seoul
  - Korea University Guro Hospital ( Site 5001), Seoul
- Spain (6):
  - Hospital Universitario Marques de Valdecilla ( Site 1602), Santander, Cantabria
  - Complexo Hospitalario Universitario de Ourense-MEDICAL ONCOLOGY ( Site 1609), Ourense, Orense
  - Hospital Universitario General de Asturias ( Site 1601), Oviedo, Principality of Asturias
  - Hospital General Universitari Vall d Hebron ( Site 1607), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 1604), Madrid
  - Hospital Virgen del Rocio ( Site 1606), Seville
- Taiwan (6):
  - Chi Mei Hospital - Liouying Branch-Clinical Trial Center ( Site 6007), Tainan, Tainan
  - Chang Gung Med Foundation. Kaohsiung Branch ( Site 6005), Kaohsiung City
  - China Medical University Hospital ( Site 6003), Taichung
  - National Cheng Kung University Hospital ( Site 6004), Tainan
  - National Taiwan University Hospital ( Site 6001), Taipei
  - Taipei Veterans General Hospital ( Site 6006), Taipei
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital ( Site 7002), Bangkok, Bangkok
  - Songklanagarind hospital ( Site 7001), Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (8):
  - Adana Medical Park Seyhan Hastanesi-Medikal Onkoloji ( Site 1714), Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 1701), Ankara
  - Memorial Ankara Hastanesi ( Site 1702), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 1715), Ankara
  - Atatürk Üniversitesi-onkoloji ( Site 1712), Erzurum
  - Acibadem Universitesi Atakent Hastanesi-Medical Oncology ( Site 1716), Istanbul
  - Istanbul Okmeydanı Egitim ve Arastirma Hastanesi ( Site 1711), Istanbul
  - Medeniyet Universitesi Tip Fakultesi ( Site 1703), Istanbul
- Ukraine (11):
  - Chernihiv Medical Center of Modern Oncology ( Site 1811), Chernihiv, Chernihiv Oblast
  - Regional Municipal Non-profit Enterprise "Bukovinian Clinical Oncology Center" ( Site 1819), Chernivtsi, Chernivetska Oblast
  - MI Kryvyi Rih Oncology Dispensary of Dnipropetrovsk Regional Council ( Site 1804), Kryviy Rih, Dnipropetrovsk Oblast
  - Kharkiv Regional Clinical Oncology Center ( Site 1812), Kharkiv, Kharkivs’ka Oblast’
  - Institute of General and Emergency Surgery n.a Zaitsev NAMS of Ukraine ( Site 1813), Kharkiv, Kharkivs’ka Oblast’
  - Communal nonprofit enterprise "Kherson Regional Oncology Dispensary" of Kherson Regional Council (, Antonivka Village, Kherson Oblast
  - SNPE National Cancer Institute ( Site 1806), Kyiv, Kyivska Oblast
  - Rivne Regional Clinical Hospital ( Site 1817), Rivne, Rivne Oblast
  - Podillya Regional Center of Oncology ( Site 1809), Vinnytsia, Vinnytsia Oblast
  - Volyn Regional Oncological Dispensary ( Site 1816), Lutsk, Volyn Oblast
  - Shalimov Institute of Surgery and Transplantation ( Site 1818), Kyiv
- United Kingdom (9):
  - Cambridge University Hospitals NHSFT ( Site 1908), Cambridge, Cambridgeshire
  - Ninewells Hospital and Medical School ( Site 1907), Dundee, Dundee City
  - Nottingham University Hospital NHS Trust ( Site 1910), Nottingham, England
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 1915), London, London, City of
  - University College London Hospitals NHS Foundation Trust ( Site 1901), London, London, City of
  - Royal Marsden NHS Foundation Trust ( Site 1905), London, London, City of
  - Royal Marsden NHS Trust. ( Site 1906), Sutton, London, City of
  - Western General Hospital ( Site 1912), Edinburgh, Midlothian
  - The Christie NHS Foundation Trust ( Site 1909), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Sun JM, Adenis A, C Enzinger P, Shah MA, Kato K, Bennouna J, Doi T, Hawk NN, Yu L, Shah S, Bhagia P, Shen L. LEAP-014: first-line lenvatinib + pembrolizumab + chemotherapy in advanced/metastatic esophageal squamous cell carcinoma. Future Oncol. 2024;20(35):2709-2721. doi: 10.2217/fon-2022-1148. Epub 2024 May 2. PMID 38695479
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26316&tenant=MT_MSD_9011